CLINICAL TRIAL: NCT04406298
Title: Safety and Efficacy of Small Frequent Paracentesis Using an Indwelling CAtheter Compared With Repeated Large Volume Paracentesis in Cirrhotic Patients With REfractory Ascites- A Randomized Controlled Trial (I-CARE)
Brief Title: Safety and Efficacy of Small Frequent Paracentesis Using an Indwelling CAtheter Compared With Repeated Large Volume Paracentesis in Cirrhotic Patients With REfractory Ascites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-29
Record Dates: First submitted 2020-05-15; First posted 2020-05-28 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-05

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small Quantity Paracentesis (Experimental): Intermittent small quantity (upto 3L per day) paracentesis through an indwelling catheter for up to 5 days.
  Interventions: Procedure: small quantity paracentesis
- Large Volume Paracentesis (Active Comparator): Large Volume Paracentesis > 5 litres
  Interventions: Procedure: Large Volume Paracentesis

INTERVENTIONS:
Procedure: small quantity paracentesis — Intermittent small quantity paracentesis (upto 3L/day) for upto 5 days
  Arms: Small Quantity Paracentesis
Procedure: Large Volume Paracentesis — Large Volume Paracentesis > 5litres
  Arms: Large Volume Paracentesis

SUMMARY:
The aim of the study is to assess the efficacy of intermittent small quantity (upto 3L per day) paracentesis through an indwelling catheter for up to 5 days in comparison with large volume paracentesis on decreasing the need for repeated paracentesis by 50 % over next 3 months. The project will be conducted at ILBS between April 2020 and March 2021. The concept of the study is to evaluate the efficacy of indwelling catheter in reducing the refilling rates of ascites by 50 % over 3 months in comparison to LVPs and also in reducing the incidence and risk of PPCD. All refractory ascites patients will be included as per inclusion and exclusion criteria, after taking informed consent from the patient or their relatives.

The expected outcomes are

Primary outcome: Proportion of cirrhotic patients with refractory ascites achieving at least 50 % reduction on need for large volume paracentesis after a short duration (5day) intermittent small quantity (up to 3L/ day) paracentesis through an indwelling catheter in comparison to a single large volume paracentesis in the next 3 months.

Secondary outcome:

1. Proportion of cirrhotic patients with refractory ascites developing P 2 . During a 30 D, 60 D and 90 D follow up, to assess between the groups

* Need for repeated paracentesis : Number assessed
* AKI : Improvement or worsening of renal functions
* Hepatic encephalopathy: Grading as per West Haven Classification
* Hyponatremia
* Diuretic tolerability : Dose and duration tolerated
* Bacterial peritonitis : Ascitic fluid neutrophil count > 250 cells/cumm
* Transplant free survival
* Risk of procedure related complications
* Changes in MELD or CTP between the groups ( Improvement vs worsening )
* Need for hospitalization between the groups

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients 18-70 yrs with refractory severe ascites with stable renal function (S.creatinine < 2 mg/dl).

Exclusion Criteria:

* CTP >12, MELD>25
* Prior or current Spontaneous Bacterial Peritonitis (SBP)
* Recurrent or current overt hepatic encephalopathy
* Serum Creatinine >2
* HVOTO (Hepatic Venous Outflow Tract Obstruction)
* Hepatic or extrahepatic malignancy
* Recent UGI bleed
* Sepsis
* Serum Sodium < 120

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-04 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of cirrhotic patients with refractory ascites achieving at least 50 % reduction on need for large volume paracentesis in both groups | 3 Months

SECONDARY OUTCOMES:
Number of participants which requires repeated paracentesis in both groups | 30 days
Number of participants which requires repeated paracentesis in both groups | 60 days
Number of participants which requires for repeated paracentesis in both groups | 90 days
Number of participants with AKI : Improvement or worsening of renal functions in both groups | 30 days
Number of participants with AKI : Improvement or worsening of renal functions in both groups | 60 days
Number of participants with AKI : Improvement or worsening of renal functions in both groups | 90 days
Number of participants with Hepatic Encephalopathy in both groups | 30 days
  Grading of Hepatic Encephalopathy will be as per West Haven Classification (Score 1 to 4) in both groups
Number of participants with Hepatic Encephalopathy in both groups | 60 days
  Grading of Hepatic Encephalopathy will be as per West Haven Classification (Score 1 to 4) in both groups
Number of participants with Hepatic Encephalopathy in both groups | 90 days
  Grading of Hepatic Encephalopathy will be as per West Haven Classification (Score 1 to 4) in both groups
Number of participants with Hyponatremia in both groups | 30 days
Number of participants with Hyponatremia in both groups | 60 days
Number of participants with Hyponatremia in both groups | 90 days
Diuretic tolerability : Dose tolerated in both groups | 30 days
Diuretic tolerability : Dose tolerated in both groups | 60 days
Diuretic tolerability : Dose tolerated in both groups | 90 days
Diuretic tolerability : Duration tolerated in both groups | 30 days
Diuretic tolerability : Duration tolerated in both groups | 60 days
Diuretic tolerability : Duration tolerated in both groups | 90 days
Bacterial peritonitis : Ascitic fluid neutrophil count > 250 cells/cumm in both groups | 30 days
Bacterial peritonitis : Ascitic fluid neutrophil count > 250 cells/cumm in both groups | 60 days
Bacterial peritonitis : Ascitic fluid neutrophil count > 250 cells/cumm in both groups | 90 days
Transplant free survival in both groups | 30 days
Transplant free survival in both groups | 60 days
Transplant free survival in both groups | 90 days
Number of participants develop adverse events associated with procedure in both groups | 30 days
Number of participants develop adverse events associated with procedure in both groups | 60 days
Number of participants develop adverse events associated with procedure in both groups | 90 days
Change in Model for End Stage Liver Disease Score in both groups | 30 days
  MELD Score ranges from 6 to 40
Change in Model for End Stage Liver Disease Score in both groups | 60 days
  MELD Score ranges from 6 to 40
Change in Model for End Stage Liver Disease Score in both groups | 90 days
  MELD Score ranges from 6 to 40
Change in CTP (Child-Turcotte-Pugh) Score in both groups | 30 days
  Child class A: < 7 points. Child class B: 7-9 points. Child class C: ≥10 points
Change in CTP (Child-Turcotte-Pugh) Score in both groups | 60 days
  Child class A: < 7 points. Child class B: 7-9 points. Child class C: ≥10 points
Change in CTP (Child-Turcotte-Pugh) Score in both groups | 90 days
  Child class A: < 7 points. Child class B: 7-9 points. Child class C: ≥10 points
Number of patients required hospitalization between the groups | 30 days
Number of patients required hospitalization between the groups | 60 days
Number of patients required hospitalization between the groups | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided